CLINICAL TRIAL: NCT05687942
Title: The REBUILD Trial: A Prospective, Multi-Center, Single Arm Study Using REBUILD for Abdominal Wall Closure
Brief Title: The REBUILD Trial: Closure of the Abdominal Wall
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AbSolutions Med Inc. (Industry)
Collaborators: Cogent Technologies Corporation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CTP-0002
Record Dates: First submitted 2023-01-08; First posted 2023-01-18 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Surgical Incision
Keywords: abdominal wall closure; hernia; laparotomy; suture tension; REBUILD
MeSH Terms: conditions — Surgical Wound; Hernia

STUDY DESIGN:
Intervention Model Description: The scientific rationale for a single-arm study is based on existing data and experience associated with current approaches for managing abdominal closure. Suture techniques and mesh have been extensively studied (Deerenberg EB, 2015) (Jairam, 2017) and several clinical publications serve as historical precedents for the 1-month endpoint (Table 2). The results of this REBUILD Study will thus exist in a broad context of outcomes, allowing significant comparisons in the absence of a concomitant control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- REBUILD (Experimental): REBUILD is an investigational medical device (bioabsorbable anchor and deployment instruments) used with third party suture to close the abdominal wall. As the suture and Anchor absorb, abdominal wall forces gradually transfer to the organizing scar, one of the tenets of successful wound tensile strength acquisition. After full absorption, no permanent material remains that would otherwise alter normal anatomy, anisotropic properties, or compliance of the abdominal wall (Deeken, 2017).
  Interventions: Device: REBUILD

INTERVENTIONS:
Device: REBUILD — 3.1.1. REBUILD is an investigational medical device provided as a sterile, single use set containing 10 suture Anchors and two non-implantable Carriers, with reusable stainless-steel instruments for deployment supplied separately.
  Other Names: REBUILD Bioabsorbable, The REBUILD System

SUMMARY:
The main objective of this clinical trial is to demonstrate the safety and efficacy of REBUILD when used to support abdominal wall closure after laparotomy. The main question it aims to answer are whether the device when used to support suture in abdominal wall closure safely maintains apposition of the abdominis rectus muscles within a pre-defined distance.

Participants will undergo standard of care laparotomy and the investigational device will be used to support the suture used to close the abdominal wall. Participants will have an MRI at 1-month after surgery to measure the distance between the abdominus rectus muscles.

DETAILED DESCRIPTION:
The REBUILD Trial (Protocol CTP-0002) is an investigational medical device study designed to demonstrate the efficacy and safety of REBUILD for abdominal wall closure (AWC). The primary evaluation period will include the first 30 days of follow up. After the 1-month endpoint evaluation period, additional follow-up at 3, 6, 12, and 24-months for post-market analysis and publication will be conducted. All adverse events will be collected and reported for the full duration of the study.

* Primary efficacy endpoint will be evaluated based on the measured distance between the rectus abdominis muscles (RAMs) by MRI at 1-month (Day 30 +14/-7 days) post-surgery (Day 0).
* Primary safety endpoint will be evaluated based on reported serious device-related adverse events through 1-month (Day 30 +14/-7 days) of follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is 22-80 years of age
2. Patient is undergoing a midline laparotomy procedure
3. Patient is able to provide written informed consent
4. Patient is able and willing to comply with all study requirements

Exclusion Criteria:

1. Patient has BMI > 40
2. Patients with available imaging measuring abdominal wall thickness < 5.7 mm or > 16.5 mm
3. Patient is scheduled for a palliative procedure or has a life expectancy of less than 12-months
4. Patient has mesh at the site of deployment
5. Patient has an ostomy within the planned midline closure site (4 cm either side of midline)
6. Patient has a CDC wound classification of Class IV
7. Patient has devitalized tissue present at the intended surgical site
8. Patient has any co-morbid conditions determined by the investigator to place them at a high risk of complications (e.g., severe cardiovascular disease, congestive heart failure NYHA Class III or IV, end-stage renal failure, liver cirrhosis, connective tissue disorder, poorly managed diabetes)
9. Patient is on any medication that the investigator determines creates a high risk for complications (e.g., antithrombotic, steroid, IV chemotherapy, immunosuppressive agent)
10. Patient has history of radiation therapy targeting the abdominal wall
11. Patient is participating in a concurrent investigational medical device study
12. Patient is pregnant or planning on becoming pregnant during the study period
13. Patient has a history of psychological condition, drug, or alcohol misuse which may interfere with their ability to be compliant with post-operative visits

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Efficacy Measure distance between the rectus abdominus muscles | Day 30 (+14/-7 days)
  The primary efficacy endpoint is a maximum distance between the RAMs at 1-month after surgery < 2.5 cm (binary outcome).
Serious device related adverse events | Day 30 (+14/-7 days)
  The primary safety endpoint is serious device-related adverse events through 1-month follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Health Care Campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No